CLINICAL TRIAL: NCT00606970
Title: Assessment of the Safety of Dietary Supplement Lactobacillus Fermented Extract in Cancer Patients Undergoing Chemotherapy
Brief Title: Safety Assessment of Lactobacillus Fermented Extract in Cancer Patients Undergoing Chemotherapy
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: FDA sent letter to IRB stating it should be done under new drug application
Sponsor: New Hope Medical Center (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Seigen Safety Trial: Cancer; WIRB Study No. 1085894; WIRB Pr. No. 20062258
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Cancer
Keywords: Chemotherapy; Breast Cancer; Colon Cancer; Lung Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Seigen Alpha EV Treatment
  Interventions: Dietary Supplement: Seigen Alpha EV
- 2 (Placebo Comparator): Identically packaged placebo packets taken 3x daily for 3 months maximum
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Seigen Alpha EV — Orally administered Seigen Alpha EV, 1 packet (6 grams)3 times daily, for maximum of 3 months. Each packet is clearly marked for breakfast, lunch, or supper. The contents are to be dissolved in water or liquid and taken orally with meal. Subjects will be required to return any unused packets to study doctor at end of each month.
  Other Names: Lactobacillus fermented extract
  Arms: Intervention group
Dietary Supplement: Placebo Comparator — Identically packaged placebo packets (each 6 grams) taken 3x daily with meals for 3 months maximum.
  Other Names: Placebo packaged identically to Seigen Alpha EV
  Arms: 2

SUMMARY:
Project: Assessment of the safety of dietary supplement lactobacillus fermented extract in cancer patients undergoing chemotherapy

Nausea and vomiting are significant causes of nutritional depletion and result in further deterioration of the physical and mental status. Support of gastrointestinal function may alleviate nausea and vomiting from chemotherapy and will not only reduce the discomfort experienced by the patient but will allow better tolerance of the treatment. This study will assess orally administered Seigen alpha EV during chemotherapy for its safety and effects on the nutritional depletion deriving from the chemotherapy. It will also look at its effect on the immune system in patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Randomization and Treatment: The subjects will be distributed in each of the three cancer categories (breast, lung, and colon), and randomized on centralized randomization lists for each of the cancer categories and assigned a unique identification number in the temporal order of recruitment. Using randomization with the minimization method, subjects will be allocated to treatment or placebo, 15 each for the treatment group or the placebo group, for a total of 30 subjects in each of the 3 cancers. This study utilizes a double-blind.

Placebo: The placebo is identical in packaging and appearance to the treatment. Identification of placebo vs. Seigen alpha EV is by unique packaging code. Patients and study doctors are blinded to the identification interpretation.

Treatment: Treatment will be for a maximum of 3 months. The dosage of the study supplement is as follows: Subjects will be instructed to take 1 packet (6 grams) 3 times daily for a total daily dosage of 3 packets (18 grams). Each packet is clearly marked for breakfast, lunch, or supper. The contents of the packet will be dissolved in water or liquid and taken orally morning, noon, and evening. Subjects will be required to return any unused packets to study doctor at the end of each month.

Assessment:

Usual clinical tests for therapeutic monitoring of usual treatment of patient will be performed.

In addition, quantitative and qualitative parameters will be measured at start of treatment and at 1, 2, and 3 months:

1. Toxicity assessments using National Cancer Institute Common Toxicity Criteria (NCI CTC): total WBC, total lymphocyte count, hemoglobin, platelet count, nausea, vomiting, diarrhea, loss of appetite, weight loss, anorexia, urticaria, fatigue, muscle weakness and headache. (Refer to Document 1 Toxicity Assessment)
2. Self-assessment of quality of life will be performed using European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 (version 3). The treating physician will summarize the patient quality of life by using the Karnofsky performance scale.
3. Additional blood test for 10 colon CA subjects (5 treatment, 5 placebo ) Molecular marker NFκB mediated signal transduction pathway genes (n=84) will be measured on 10 subjects with colon cancer. A sample of no less than 5 ml using PAXgene Blood RNA Tubes (Qiagen, Cat. No. 762115) will be collected from each subject. Shipment overnight on at least 10 lbs of ice block (blue or wet) to SuperArray Bioscience in Frederick, MD 21704.

Baseline and repeated at one, two and three months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects have given written informed consent prior to participation
* They must have a life expectancy of greater than 6 months
* They must have biopsy confirmed primary breast, colon or lung cancer
* They are receiving standard chemotherapy in accordance with American Society Clinical Oncology (ASCO) standards and have at least one month remaining in their chemotherapy course
* They must have an Eastern Cooperative Oncology Group (ECOG) performance status < 2 and are being treated as outpatients.
* Subjects must be between the ages of 18 to 75 years of age.
* Subjects must be able to communicate in English.

Exclusion Criteria:

* Have received radiotherapy within the last 4 weeks
* Have acute gastrointestinal problems e.g. acute gastrointestinal infection, gastric or duodenal ulcer, history of bowel obstruction, diverticulitis, Crohn's disease, ulcerative colitis, or chronic diarrhea
* Presence or clinical evidence of CNS metastases
* Receiving corticosteroids
* Have severe concomitant disease
* Have severe dysphagia, esophagitis or xerostoma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in self-rated symptoms and assessed signs | 3 months

SECONDARY OUTCOMES:
Affect on treatment results | 3 months maximum

CONTACTS AND LOCATIONS:
Overall Officials: Ed Fujimoto, PhD, Study Director — New Hope Medical Center